CLINICAL TRIAL: NCT01589211
Title: Brief Intervention Study for Quitting Smoking
Acronym: BISQUITS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Necessary number of participants not achieved and high drop out rate
Sponsor: Heidelberg University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Felix JF Herth, Dr. med. Alexander Rupp, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WS899101
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Smoking; Tobacco Use Cessation; Smoking Cessation
Keywords: smoking; cessation; intervention; brief
MeSH Terms: conditions — Smoking; Tobacco Use Cessation; Smoking Cessation | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief advice (Active Comparator): A brief advice to stop smoking of about 10 min accompanied with self-help material
  Interventions: Behavioral: Brief advice
- Compact cessation course (Experimental): Cessation intervention of 2 x 120 min in a group setting
  Interventions: Behavioral: Compact cessation course
- Standard cessation course (Active Comparator): Cessation course in a group setting over 6 dates
  Interventions: Behavioral: Standard cessation course

INTERVENTIONS:
Behavioral: Brief advice — Brief advice of about 10 min accompanied by self-help material
  Arms: Brief advice
Behavioral: Compact cessation course — Compact cessation course on the basis of Motivational Interviewing (MI) and Cognitive Behavioural Therapy (CBT). Group setting. 2 x 120 min.
  Arms: Compact cessation course
Behavioral: Standard cessation course — Cessation course over 6 dates. Group setting.
  Arms: Standard cessation course

SUMMARY:
To investigate the effectiveness of a smoking cessation intervention of two sessions (120 min at a time) in a group setting on the basis of Motivational Interviewing (MI) and important elements of Cognitive Behavioural Therapy (CBT). According to national and international guidelines patients are advised to quit and pharmacologically supported with one of the established first line smoking cessation treatments.

DETAILED DESCRIPTION:
The study design is multicentric, prospective, randomized and controlled. The study is taking place in cooperation with smoking clinics of 5 centres in Germany (Heidelberg, Stuttgart, Munich, Chemnitz, Berlin). A total number of 800 smokers is calculated to participate in the study. After enrollment participants are randomized in one of the three intervention groups: (A) "Advice only", (B) "Brief intervention", (C) "Intensive therapy". The follow up includes a telephone interview 3 months after the last intervention, and two visits at the smoking clinics after 6 and 12 months with biochemical validation of the smoking status by measurement of the exhaled carbon monoxide and the concentration of cotinine in an urine sample respectively. The primary endpoint is the continuous abstinence rate after 12 months. Several secondary endpoints are determined amongst others the continuous abstinence rate after 6 months, point prevalence cessation rates after 6 and 12 months, life quality, weight gain, predictors of a successful cessation attempt.

ELIGIBILITY:
Inclusion Criteria:

* Smoker
* Age > 18 years
* Motivation to quit smoking

Exclusion Criteria:

* severe somatic comorbidity or reduced life expectancy
* severe episode of a psychiatric disease
* reduced cognitive ability
* abuse of alcohol or illicit drugs
* other reasons at the discretion of responsible local study tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2011-12-16 (Actual); Primary Completion 2013-04-11 (Actual); Study Completion 2013-04-11 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence rate | 12 months
  Biochemical validation by measurement of urine cotinine levels

SECONDARY OUTCOMES:
Continuous abstinence rate | 6 months
Time point abstinence rate | 6 and 12 months
Quality of life (SF36 short form) | 0, 6 and 12 months
  Quality of life
Depression | 0, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rupp, Dr., Principal Investigator — Heidelberg University; Michael Kreuter, PD Dr., Study Chair — Heidelberg University; Felix JF Herth, Prof., Study Director — Heidelberg University
Locations (5):
- Germany (5):
  - Thoraxklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Pneumologische Praxis im Zentrum (former: Zentrum für Tabakentwöhnung Stuttgart), Stuttgart, Baden-Wurttemberg
  - Klinikum der Universität München - Klinik für Psychiatrie und Psychotherapie, Munich, Bavaria
  - Technische Universität Chemnitz - Institut für Psychologie, Chemnitz, Saxony
  - Institut für Raucherberatung und Tabakentwöhnung am Gemeinsschaftskrankenhaus Havelhöhe, Berlin

REFERENCES:
- [Background] Rupp A, Blank J, Ehmann M, Pousset R, Mühlig S, Sehl A, Fuchs S, Rüther T, Linhardt A, Grah C, Kreuter M. Basic data of the Brief Intervention Study for Quitting Smoking (BISQUITS). Pneumologie. 2014; 68 - P106 DOI: 10.1055/s-0034-1367889